CLINICAL TRIAL: NCT01912859
Title: Next Steps: a Community-led Solution to Sustaining Healthy Behaviors in Families Addressing Childhood Obesity
Brief Title: Next Steps: a Community-led Solution to Address Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other); The Family Partnership, Minneapolis (Unknown); Community Leaders, Minneapolis, Richfield (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1303S29343
Record Dates: First submitted 2013-07-18; First posted 2013-07-31 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition/physical activity intervention (Experimental): The intervention, Next Steps, comprises a network of community-led health maintenance programs offered to graduates of an initial intensive obesity course. These health maintenance programs will aim to help participants maintain and improve healthful behaviors and body mass indices.
  Interventions: Behavioral: Nutrition/physical activity intervention
- Usual care (No Intervention): Participants in the "No Intervention" arm will not have access to the Next Steps programs and will receive only usual care through their health care clinic.

INTERVENTIONS:
Behavioral: Nutrition/physical activity intervention — Nutrition/physical activity intervention
  Arms: Nutrition/physical activity intervention

SUMMARY:
The purpose of Next Steps pilot intervention is to develop and test a new program designed to help low-income multiethnic families with overweight or obese children achieve long-term maintenance of healthful behaviors following completion of Hennepin County Medical Center's (HCMC) 16-week intensive obesity management course (Taking Steps Together (TST)).

DETAILED DESCRIPTION:
Next Steps is a community based pilot intervention study conducted in collaboration between community leaders, the University of Minnesota, Hennepin County Medical Center (HCMC) and The Family Partnership. The study collaborators will develop and test a new program designed to help low-income multiethnic families with overweight or obese children achieve long-term maintenance of healthful behaviors following completion of HCMC's 16-week intensive obesity management course (Taking Steps Together (TST)). Next Steps, the focus of this study, will comprise a network of parent-led, community-based health maintenance programs that will be offered to TST graduate families.

Project Aims:

Aim 1: Establish a core parent leadership group and health maintenance program network that is self-sustaining and can serve the community for years to come.

Aim 2: Test the feasibility, acceptability and sustainability of the Next Steps programs.

Aim 3: Assess the impact of the Next Steps programs on helping participant families sustain or improve healthful behaviors and achieve or maintain healthy body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Families that are graduates of the Taking Step Together program.
* Families with at least one overweight or obese child between the ages of 7-17.
* Family members of all ages who have graduated from the Taking Steps Together program will be included in the study.

Exclusion Criteria:

* Families who are not graduates of the Taking Steps Together program.
* Families who do not have one child that is between the ages of 7-17 and who is overweight or obese

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maintain or lower body mass index | up to 4 months
  Body mass index.
Frequency and intensity of physical activity | up to 4 months
  Frequency and intensity of physical activity
Frequency of intake of healthful foods and reduction of unhealthful foods; | up to 4 months
  Frequency of intake of healthful foods and reduction of unhealthful foods;

CONTACTS AND LOCATIONS:
Overall Officials: Chrisa Arcan, PhD, Principal Investigator — University of Minnesota; John D Anderson, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis; Maria Galvan, Principal Investigator — Community Leader; Natividad Contreras, Principal Investigator — Community Leader; Aurolivia Reyes, Principal Investigator — Community Leader